CLINICAL TRIAL: NCT06568393
Title: The Effect of Calisthenic Exercises on Quality of Life in Post-Covid Syndrome: A Randomized Controlled Trial
Brief Title: Effectiveness of Calisthenic Exercises in Post-Covid Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Alper Percin, Asst. Prof., Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AP0007
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Quality of Life
Keywords: Post-COVID Condition; Long COVID; Life Quality; Exercise Training
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: The study was conducted in 2 groups, one intervention and one control group.
Who Masked: Outcomes Assessor
Masking Description: The assessment was completed by a another therapist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calisthenic (Experimental): In this group, calisthenic exercises were performed by a therapist with face to face and it was taken for 8 weeks.
  Interventions: Other: Calisthenic exercise
- Home exercise (Active Comparator): In this group, a home exercise programme of calisthenic exercises was prepared and shown to the participants with visuals and they were asked to perform this exercise programme for 8 weeks.
  Interventions: Other: Calisthenic exercise

INTERVENTIONS:
Other: Calisthenic exercise — Calisthenic exercise program was included: jumping jack, burpee, mountain climber, squat thrust, squat, squat jump, split and alternate exercises.

SUMMARY:
Post-Covid syndrome is known as the appearance of some symptoms for 12 weeks or more after Covid-19 infection, affecting the patient's quality of life. The wide range of symptoms that occur after post-Covid syndrome has led to the development of different interventions. In this study, we tried to measure changes in quality of life in people with post-covid syndrome as a result of using calisthenics with therapists and home exercise. Quality of life scale scores were compared before and after an 8-weeks exercise intervention.

DETAILED DESCRIPTION:
In this study, a quantitative approach with a pre-test-post-test design was applied to compare the effect of calisthenic exercises on quality of life in individuals with post-covid syndrome in the form of a therapist-guided and home exercise programme. Participants signed an informed consent form before inclusion in the study and the details of the study were clearly explained. At baseline, age, gender, height, weight, symptoms and duration of symptoms were recorded. Quality of life data were recorded with the EQ-5D-3L questionnaire at baseline and 8 weeks after the exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

* To be 18 years of age or older, previous having Covid-19 infection, 12 weeks or more of post-covid symptoms.

Exclusion Criteria:

* The presence of acute viral or bacterial infection, having been previously diagnosed with a rheumatic, neurological, metabolic or oncological disease, having undergone any surgical procedure after musculoskeletal injury, use of intra-articular prosthesis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
EQ-5D-3L (European Quality of Life 5 Dimensions 3 Level Version) | Baseline of the study
  Depending on the answers given in this questionnaire, 1 - 3 points are assigned, while a low score indicates a healthy state, a high score indicates a problem that reduces the quality of life. In the second part of the questionnaire, there is a part where a score between 0-100 is asked to explain the state of being healthy today, in this part, low scores indicate that there are health problems and high scores define the state of being healthy.

CONTACTS AND LOCATIONS:
Overall Officials: Alper Percin, Asst. Prof., Principal Investigator — Bahçeşehir University
Locations (1):
- Igdır University, Iğdır, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Domaszewska K, Boraczynski M, Tang YY, Gronek J, Wochna K, Boraczynski T, Wielinski D, Gronek P. Protective Effects of Exercise Become Especially Important for the Aging Immune System in The Covid-19 Era. Aging Dis. 2022 Feb 1;13(1):129-143. doi: 10.14336/AD.2021.1219. eCollection 2022 Feb. PMID 35111366
- [Background] Muniswamy P, Gorhe V, Parashivakumar L, Chandrasekaran B. Short-term effects of a social media-based intervention on the physical and mental health of remotely working young software professionals: A randomised controlled trial. Appl Psychol Health Well Being. 2022 May;14(2):537-554. doi: 10.1111/aphw.12318. Epub 2021 Nov 8. PMID 34750975
- [Background] Tekin F, Cetisli-Korkmaz N. Effectiveness of a Telerehabilitative Home Exercise Program on Elder Adults' Physical Performance, Depression and Fear of Falling. Percept Mot Skills. 2022 Jun;129(3):714-730. doi: 10.1177/00315125221087026. Epub 2022 Apr 11. PMID 35404709